CLINICAL TRIAL: NCT01868438
Title: Phase 1, Open-label, Cross-over Study to Investigate the Relative Bioavailability of Pyramax (Pyronaridine-artesunate) in Tablet and Granule Formulations, in Healthy Volunteers
Brief Title: Relative Bioavailability of Pyronaridine-artesunate in Tablet and Granule Formulations in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Medicines for Malaria Venture (Other)
Collaborators: Shin Poong Pharmaceutical Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SP-C-017-12
Record Dates: First submitted 2013-05-30; First posted 2013-06-04 (Estimated); Results first posted 2023-12-18 (Actual); Last update posted 2023-12-18 (Actual); Status verified 2023-12

CONDITIONS: Malaria
Keywords: Pyronaridine artesunate tablet; Pyronaridine artesunate granules; Pyramax tablet; Pyramax granules; Bioavailability; artemisinin based combination therapy (ACT)
MeSH Terms: conditions — Malaria | interventions — pyronaridine tetraphosphate, artesunate drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pyronaridine-artesunate granules (Period 1) (Active Comparator): Period 1: single administration of pyronaridine-artesunate granules: total dose 540mg pyronaridine + 180mg artesunate.
  Period 2: cross-over to single administration of pyronaridine-artesunate tablets: total dose 540mg pyronaridine + 180mg artesunate.
  Interventions: Drug: Pyronaridine-artesunate granules; Drug: Pyronaridine-artesunate tablets
- Pyronaridine-artesunate tablets (Period1) (Active Comparator): Period 1: single administration of pyronaridine-artesunate tablets: total dose 540mg pyronaridine + 180mg artesunate.
  Period 2: cross-over to single administration of pyronaridine-artesunate granules: total dose 540mg pyronaridine + 180mg artesunate.
  Interventions: Drug: Pyronaridine-artesunate granules; Drug: Pyronaridine-artesunate tablets

INTERVENTIONS:
Drug: Pyronaridine-artesunate granules
  Other Names: Pyramax granules; PA granules
Drug: Pyronaridine-artesunate tablets
  Other Names: Pyramax tablets; PA tablets

SUMMARY:
The primary objective of this study is to compare the bioavailability of two formulations (tablets and granules for dispersion) of the antimalarial drug pyronaridine-artesunate [3:1] (Pyramax, PA) in healthy adults. The secondary objective is to compare the safety of the two PA formulations and liver function test changes following the first and second administrations.

DETAILED DESCRIPTION:
This is a Phase I, single centre, open-label, randomised, two-way cross-over study in healthy volunteers to compare the bioavailability of two formulations of pyronaridine-artesunate, in tablet and in granule formulation. The study population will include 60 healthy volunteers, comprising male and female adults aged 20 to 45 years inclusive.

The volunteers will be randomised equally on Day -1 to one of two sequences: Sequence 1 (tablets in Period 1, granules in Period 2), or Sequence 2 (granules in Period 1, tablets in Period 2). The periods will be separated by a 60-day wash-out period. Each of the two pyronaridine-artesunate formulations will be administered as a single dose of either 180:60 mg pyronaridine-artesunate tablets (3 tablets) or 60:20 mg pyronaridine-artesunate granules (9 sachets). The total dose of each formulation administered is 540:180 mg pyronaridine-artesunate.

The study duration from the first study drug administration (Day 1) through to the last follow-up will be approximately 103 days. Screening is to be performed within 28 days before Day 1. Adverse events will be monitored throughout the study (and to resolution if necessary) to assess the general safety and tolerability of the treatments.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male and/or female subjects between the ages of 20 and 45 years, inclusive. (Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12-lead ECG and clinical laboratory tests)
* Weight between 50 kg and 80 kg and Body Mass Index (BMI) calculated using Quetelet's Index - weight(kg)/height (m2) between 18.5 to 27 kg/m2;
* An informed consent document signed and dated by the subject (prior to screening and any study activities, including discontinuation of any prohibited medications)
* Strictly normal values of alanine aminotransferase(ALT), aspartate aminotransferase (AST), and bilirubin, and normal or abnormal but clinically insignificant results of the other blood and urine laboratory parameters at screening.
* Female subjects of non-childbearing potential [i.e., physiologically incapable of becoming pregnant, including any female who was post-menopausal (i.e., one year without menses) or who has undergone sterilization (via hysterectomy or bilateral tubal ligation)]
* Female subjects of childbearing potential with a negative urine pregnancy test at screening, and a negative pregnancy blood test on admission, and who :

  * agree to double barrier method of contraception for 4 weeks before first study drug administration and throughout the entire study follow up period, or
  * whose partner has undergone vasectomy and has been negative for sperm for at least 6 months
* Subjects who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

* Known history or evidence of clinically significant disorders such as cardiovascular (including arrhythmia, acute corrected QT interval (QTc) greater or equal to 450 milliseconds), respiratory (including active tuberculosis), hepatic, renal, gastrointestinal, immunological (including active HIV-AIDS), neurological (including auditory), endocrine, infectious, malignancy, psychiatric or other abnormality (including head trauma)
* Known history of hypersensitivity, allergic or adverse reactions to pyronaridine or artesunate or other artemisinins
* Known active Hepatitis A IgM (HAV-IgM), Hepatitis B surface antigen (HBsAg) or Hepatitis C antibody (HCV Ab)
* Seropositive HIV antibody, seropositive syphilis [Syphilis reagin test (+)]
* Previous exposure to pyronaridine-artesunate (Pyramax)
* Present or recent history (last two years) of tobacco abuse (≥10 cigarettes/day)
* Known or suspected alcohol abuse or illicit drug use up to 5 years before the study start or positive findings on urine drug screen
* Intake of alcoholic beverages or caffeine-containing food or beverages, such as coffee, tea, chocolate, or cola, 48 hours before study drug administration
* Intake of grapefruit, Seville oranges or products containing these from 72 hours before the start of study drug administration
* Gilbert's disease
* Use of over-the-counter (OTC) medications, including vitamins, analgesics, antipyretics or antacids within 7 days before study drug administration
* Use of prescription medications within 14 days before the start of study drug administration or required chronic use of any prescription medication
* Use of enzyme-altering agents (e.g. barbiturates, phenothiazines, cimetidine, etc.) within 30 days before the start of study drug administration
* Plasma donation within 60 days before the start of study drug administration
* Blood donation of 500 mL or more within 60 days before the start of study drug administration
* Participation AND having had drug administration in any other clinical study within the 60 days before start of study drug administration

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2013-05; Primary Completion 2013-10 (Actual); Study Completion 2014-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Dept. of Clinical Pharmacology and Therapeutics, Asan Medical Center, Univ. of Ulsan, Seoul, South Korea

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 30 Volunteers were recruited to Sequence 1 and 30 to Sequence 2 (60 total). Since this is a crossover study from tablets to granules (Sequence 1) or vice versa (Sequence 2), overall there is a planned 60 volunteers taking tablets and 60 volunteers taking granules.
Groups:
- Pyronaridine-artesunate Tablets First, Then Pyronaridine-artesunate Granules: Participants first received a single administration of 3 180:60 mg pyronaridine-artesunate tablets. After a washout period of 60-days, they then received a single administration of 9 sachets of 60:20 mg pyronaridine-artesunate granules. Total doses for both formulations were 540mg pyronaridine + 180mg artesunate.
- Pyronaridine-artesunate Granules First, Then Pyronaridine-artesunate Tablets: Participants first received a single administration of 9 sachets of 60:20 mg pyronaridine-artesunate granules. of. After a washout period of 60-days, they then received a single administration of 3 180:60 mg pyronaridine-artesunate tablets. Total doses for both formulations were 540mg pyronaridine + 180mg artesunate.
Period: First Intervention
Arm/Group | Pyronaridine-artesunate Tablets First, Then Pyronaridine-artesunate Granules | Pyronaridine-artesunate Granules First, Then Pyronaridine-artesunate Tablets
Started | 30 | 30
Completed | 23 | 25
Not Completed | 7 | 5
Not completed — Withdrawal by Subject | 5 | 1
Not completed — Lost to Follow-up | 2 | 3
Not completed — Meeting the non-redosing criteria | 0 | 1
Period: Second Intervention
Arm/Group | Pyronaridine-artesunate Tablets First, Then Pyronaridine-artesunate Granules | Pyronaridine-artesunate Granules First, Then Pyronaridine-artesunate Tablets
Started | 23 | 25
Completed | 20 | 22
Not Completed | 3 | 3
Not completed — Adverse Event | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- All Volunteers Enrolled: Includes both tablets and granules groups
Arm/Group | All Volunteers Enrolled
Number analyzed (Participants) | 60
Age, Customized [Count of Participants; unit: Participants]
  20-24 years | 33
  25-29 years | 18
  30-39 years | 8
  40-45 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 58
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Korean | 60
BMI [Mean (Standard Deviation); unit: kg/m^2] | 22.78 (1.60)

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve From Hour 0 to the Last Sampling Point (AUC 0-t) for Pyronaridine and Dihydroartemisinin (DHA)
Description: Pharmacokinetic blood sampling for first or second intervention dose
Time Frame: First intervention: Day 1 pre-dose to Day 43 visit (D1, 2, 3, 4, 6, 8, 15, 22, 29, 36, 43) ; second intervention: Day 61 pre-dose to Day 103 visit (D61, 62, 63, 64, 66, 68, 75, 82, 89, 96, 103)
Population: Number analyzed includes only subjects completing both periods with estimable parameters.
Measure: Mean (Standard Deviation); unit: ng*h/ml
Groups:
- Total Receiving Pyronaridine-artesunate Tablets: Sequence 1: period 1 single administration of pyronaridine-artesunate tablets: total dose 540mg pyronaridine + 180mg artesunate.
  Sequence 2: period 2 cross-over to single administration of pyronaridine-artesunate tablets: total dose 540mg pyronaridine + 180mg artesunate.
- Total Receiving Pyronaridine-artesunate Granules: Sequence 2: period 1 single administration of pyronaridine-artesunate granules: total dose 540mg pyronaridine + 180mg artesunate.
  Sequence 1: period 2 cross-over to single administration of pyronaridine-artesunate granules: total dose 540mg pyronaridine + 180mg artesunate.
Arm/Group | Total Receiving Pyronaridine-artesunate Tablets | Total Receiving Pyronaridine-artesunate Granules
Number analyzed (Participants) | 42 | 42
ng*h/ml
  AUC 0-t pyronaridine: number analyzed (Participants) | 26 | 26
  AUC 0-t pyronaridine | 11640 (4344) | 11324 (3927)
  AUC 0-t DHA | 1119 (364) | 829 (328)

2. Secondary Outcome: Tmax and Terminal Half Life for Pyronaridine, Artesunate and DHA
Description: Pharmacokinetic blood sampling for first or second intervention dose
Time Frame: as for outcome 1
Population: Number analyzed includes only subjects completing both periods with estimable parameters.
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Total Receiving Pyronaridine-artesunate Tablets | Total Receiving Pyronaridine-artesunate Granules
Number analyzed (Participants) | 42 | 42
hours
  Tmax pyronaridine | 2.1 (2) | 1.7 (1.6)
  Half-life pyronaridine: number analyzed (Participants) | 26 | 26
  Half-life pyronaridine | 639 (262.2) | 591.8 (372.9)
  Tmax artesunate | 0.98 (0.544) | 1.52 (0.921)
  Half-life artesunate: number analyzed (Participants) | 6 | 6
  Half-life artesunate | 0.33 (0.0852) | 0.71 (0.112)
  Tmax DHA | 1.46 (0.69) | 2.26 (0.871)
  Half-life DHA: number analyzed (Participants) | 41 | 41
  Half-life DHA | 1.50 (0.713) | 1.43 (0.718)

3. Secondary Outcome: Safety Evaluation - Summary of Adverse Events
Time Frame: End of study (Day 103)
Measure: Count of Participants; unit: Participants
Arm/Group | Total Receiving Pyronaridine-artesunate Tablets | Total Receiving Pyronaridine-artesunate Granules
Number analyzed (Participants) | 55 | 53
Participants
  Adverse event before treatment | 2 | 0
  Treatment-emergent adverse event | 22 | 23
  Treatment-related adverse event | 14 | 14
  Serious adverse event | 0 | 0
  Serious adverse drug reaction | 0 | 0
  Adverse event leading to discontinuation | 3 | 3

ADVERSE EVENTS:
Time Frame: 103 days (end of study). All adverse events (AEs) were to be monitored up to resolution or if at the end of the study until <Grade 1 according to the World Health Organization (WHO) toxicity scale. Any serious AE (SAE) was to be monitored up to resolution or until no new medical information was expected.
Arm/Group | Total Receiving Pyronaridine-artesunate Tablets | Total Receiving Pyronaridine-artesunate Granules
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/53
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/53
Other Adverse Events (participants affected / at risk) | 22/55 | 23/53
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Total Receiving Pyronaridine-artesunate Tablets (N=55) | Total Receiving Pyronaridine-artesunate Granules (N=53)
Nausea (Gastrointestinal disorders) | 4 (4) | 6 (6)
Diarrhoea (Gastrointestinal disorders) | 2 (3) | 6 (6)
Vomiting (Gastrointestinal disorders) | 3 (3) | 3 (3)
Abdominal discomfort (Gastrointestinal disorders) | 2 (2) | 3 (4)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 2 (2) | 5 (5)
Neutrophil count decreased (Investigations) | 3 (4) | 3 (3)
Blood bilrubin increased (Investigations) | 1 (1) | 1 (1)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 1 (1)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Rhinorroea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 4 (7) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 2 (3) | 1 (1)
Hypercalcaemia (Metabolism and nutrition disorders) | 1 (3) | 0 (0)
Pyrexia (General disorders) | 2 (2) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1)
Feeling hot (General disorders) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 1 (1) | 1 (1)
Hordeolum (Infections and infestations) | 1 (1) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Xanthopsia (Eye disorders) | 0 (0) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No